CLINICAL TRIAL: NCT07313696
Title: Picture This: Learning to Focus and Savor With a Smartphone
Brief Title: Picture This: Bringing Joy Into Focus and Developing Healthy Habits of Mind
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Clark University (Other); John Templeton Foundation (Other)
Responsible Party: Principal Investigator, Laura Mckee, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H26061; ID# 43893 (Other Grant/Funding Number: John Templeton Foundation)
Record Dates: First submitted 2025-11-20; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: College Student Mental Health; Mindfulness; Positive Emotions; Savoring; Intervention Study
Keywords: positive psychology; intervention; photography; savoring; mindfulness; well-being
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Picture This! (Experimental): 1. Take 2 or more photographs each day for 21 days of something that elicits positive emotion
  2. When taking the photograph, notice: 1) how your body feels physically, 2) what thoughts are going through your mind, 3) what emotions you are experiencing.
  3. Save these photographs on your phone. Upload them to the study drive.
  4. Each evening for 21 days, take 10 minutes to review the photographs you took during the course of the day. Review the photos you took as a part of the study.
  5. Complete nightly savoring exercises online while reviewing photos taken during the day and answer questions about well-being
  6. Complete weekly brief questionnaire about well-being
  7. Complete pre and post assessments, prior to and at the end of the 21 days
  Interventions: Behavioral: Attentional focus on positive emotion via photography
- Picture This! Plus Social Sharing (Experimental): 1. Take 2 or more photographs each day for 21 days of something that elicits positive emotion
  2. When taking the photograph, notice: 1) how your body feels physically, 2) what thoughts are going through your mind, 3) what emotions you are experiencing.
  3. Save these photographs on your phone. Upload them to the study drive.
  4. Each evening for 21 days, take 10 minutes to review the photographs you took during the course of the day. Review the photos you took as a part of the study.
  5. Complete nightly savoring exercises online while reviewing photos taken during the day and answer questions about well-being
  6. Share your photos with a friend/family member each week. Complete questionnaire about sharing experience and weekly brief questionnaire about well-being
  7. Complete pre and post assessments, prior to and at the end of the 21 days
  Interventions: Behavioral: Attentional focus on positive emotion via photography; Behavioral: Social Sharing
- Document This! (Placebo Comparator): 1. Take 2 or more photographs each day for 21 days of your "day-in-the-life"
  2. When taking the photograph, notice: 1) how your body feels physically, 2) what thoughts are going through your mind, 3) what emotions you are experiencing.
  3. Save these photographs on your phone. Upload them to the study drive.
  4. Each evening for 21 days, take 10 minutes to review the photographs you took during the course of the day. Review the photos you took as a part of the study.
  5. Complete nightly savoring exercises online while reviewing photos taken during the day and answer questions about well-being
  6. Complete weekly brief questionnaire about well-being
  7. Complete pre and post assessments, prior to and at the end of the 21 days
  Interventions: Behavioral: Taking Photographs of daily life events and moments
- No Photo Control (No Intervention): 1. Each evening for 21 days, answer questions about well-being
  2. Complete weekly brief questionnaire about well-being
  3. Complete pre and post assessments, prior to and at the end of the 21 days

INTERVENTIONS:
Behavioral: Attentional focus on positive emotion via photography — The current project aims aim to test a set of exercises using Smartphones with college and graduate students designed to retrain attention toward moments/events/people that elicit positive emotions, encourage the savoring of such moments, increase social connectedness, and in turn, decrease depressive symptoms.
  Other Names: savoring; mindfulness
  Arms: Picture This!; Picture This! Plus Social Sharing
Behavioral: Social Sharing — For individuals in the social sharing condition, participants were instructed to share their photos for the study each week with a friend or family member of their choice. They were provided a script to help them with the social sharing, if needed.
  Arms: Picture This! Plus Social Sharing
Behavioral: Taking Photographs of daily life events and moments — The individuals in the Document This condition will take daily photographs of moments in their lives for 21 days. They are not directed to focus on taking photos that elicit positive affect as the individuals in PT and PTPSS are. They are asked to review their photos each evening and answer questions about them.
  Arms: Document This!

SUMMARY:
The goal of this clinical trial is to test whether photography-based, smartphone exercises can increase well-being and reduce depressive symptoms in college and graduate students. The main questions it aims to answer are:

Can savoring and/or social sharing of positive experiences via smartphone photography improve emotional well-being? Does attentional retraining toward positive stimuli reduce depressive symptoms?

Researchers compared:

Picture This! (21 days of taking daily photos of things that elicited a positive emotion, savoring the moment, and reviewing the photos at the end of each day) Picture This! Plus Social Sharing (21 days taking daily photos of things that elicited a positive emotion, savoring the moment, and reviewing the photos at the end of each day + sharing photos each week with a friend/family member) Document This! (21 days of taking "day in the life" photos each day and reviewing them each evening) Passive control group (21 days without instructions to take photos)

To see if the positive emotion-focused intervention conditions (Picture This! and Picture This! Plus Social Sharing) outperformed neutral (Document This!0 or no-photo conditions in improving psychological health.

Participants were:

Randomly assigned to one of four groups. Asked to complete baseline and follow-up questionnaires and computer tasks.

Three active conditions:

Take 2+ photos daily for 3 weeks. Upload photos to a secure drive. Complete nightly savoring exercises and surveys. (Social Sharing group only) Share photos weekly with a friend/family member.

All participants completed weekly surveys and a final lab visit with follow-up assessments.

DETAILED DESCRIPTION:
The proposed intervention draws primarily from two paradigms, positive psychology interventions (PPI) and cognitive bias modification (CBI), and marries components of each into a technology-enhanced program designed to increase global well-being and decrease social isolation and depressive symptoms among college students. Although both intervention paradigms are in relatively early stages of investigation, they have garnered an impressive amount of empirical support indicating their success with regard to increasing psychological health. While they have grown out of very different traditions and theoretical cloths, both approaches also aim to uplift individuals who are languishing rather than flourishing and provide behavioral, cognitive, and attentional tools to increase the experience of positive emotion.

Although they come in various forms ranging from the intentional practice of positive thinking to writing letters of gratitude and increasing social interactions, all positive psychology interventions (PPIs) utilize practices, tools, and exercises to cultivate or increase the participant's sense of subjective well-being. They are, by definition, strengths-based and so do not necessarily intend to address deficits or heal pathology; rather, they are designed to optimize, to build, and to elevate. Recently, PPIs have been utilized with participants suffering from depression. While this application may at first blush seem at odds with the definition, a closer look provides clarity. Depression is characterized not only by high levels of negative affect but also low levels of positive affect. Research to date indicates that increased positive emotion in depressed individuals is beneficial with regard to "increased broad-minded coping,", resilience from negative emotions, and even in preventing relapse. Accordingly, such interventions are a natural fit for depression. A recent meta-analysis suggests that PPIs are superior to control or comparison groups in enhancing well being and in addressing depressive symptoms; however, PPIs may be relatively more successful for depressed participants and participants who self-select into the interventions.

Cognitive models of depression have long posited that individuals suffering from affective disorders (namely, Major Depressive Disorder) show information processing deficits that include increased attention to negatively-valenced cues. For example, when presented with both sad and neutral faces, subjects diagnosed with MDD selectively attended to the sad face, whereas control subjects divided attention between the sad and neutral faces. More recent work indicates that dysphoric individuals lack a protective bias toward positive stimuli and that they have difficulty disengaging from "mood-congruent (i.e., sad, negative)" stimuli. There is also some evidence that depressed individuals may be more likely to interpret ambiguous stimuli as threatening. Recently, researchers have tested cognitive bias modification interventions (CBI), which are designed explicitly to modify dysfunctional patterns of information processing including both attentional and interpretation biases. In their meta-analysis of 45 CBM studies, one research group found, overall, a medium effect size for the CBMs on cognitive biases and a small, but significant, effect on anxiety and depressive symptoms before the data was corrected for publication bias. Although the effects were no longer significant after correction for publication bias, the authors report a larger and more robust (while still insignificant) effect for CBMs when measured in the context of a stressor, giving credence to the diathesis-stress cognitive paradigm. They also noted that interpretational biases were impacted relatively more than attentional biases by the intervention manipulation, and anxiety symptoms relatively more than depressive symptoms.

Building upon these two disparate bodies of research, the current project aims aim to test a set of exercises using Smartphones with college and graduate students designed to retrain attention toward moments/events/people that elicit positive emotions, encourage the savoring of such moments, increase social connectedness, and in turn, decrease depressive symptoms. The aims will be achieved by recruiting college/university/graduate students who provide consent to participate in a randomized trial of the intervention and who will be randomly be assigned to 1 of 4 conditions.

1. Those participants who are randomized to the active Picture This! savoring condition will be asked to use their Smartphones to take at least two photographs each day for 3 weeks of something that brings them joy or peace and to upload their pictures daily to a drive accessed by study staff (instructions for each condition may be found in Appendix A). Each evening, they will be directed to complete an online exercise in which they review the photograph(s) taken that day. They are also asked to complete several questions via an internet survey.
2. Participants randomized to the Picture This! Plus Social Sharing will do everything as described for the Picture This! group. In addition, each week, they will be directed to share the photos they took during the prior week with a friend or family member (see script provided in Appendix B).
3. Those participants who are randomized to the active control condition (Document This!) will also be asked to take 2 photographs each day using a Smartphone and to upload their pictures daily to a drive accessed by study staff. Rather than focusing on and capturing a photo of stimuli that evokes positive emotion, however, they will be directed to take pictures of things in their lives or surroundings that are representative of a "day in the life". Like the participants in the Picture This! and Picture This! Plus Social Sharing Groups, they will also be asked to complete an online exercise each evening in which they review their documentary photos each evening and also asked to complete a series of questions via an internet survey.
4. Finally, participants randomized to the passive control group will NOT be directed to take any pictures during the 3 week intervention period.

All research participants in all 4 groups will be asked to complete a weekly online survey asking about whether they shared the pictures they took as a part of the study or as a part of their regular life (see Appendix F).

At the end of the intervention, all subjects will be provided a list of local mental health resources and will also be provided with the instructions for all 3 picture taking conditions (should they wish to implement any of the other exercises on their own time).

ELIGIBILITY:
Inclusion Criteria:

* College, university, or grad student in urban area where data collection was taking place
* 18 years old or older
* daily access to a Smartphone with a camera
* daily access to the internet and active email address
* interest in the study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2015-05-15 (Actual); Study Completion 2015-05-15 (Actual)

PRIMARY OUTCOMES:
Mean level change from baseline to study completion in depressive symptoms for individuals in the PT and PTPSS intervention groups | from baseline to study completion (approximately 21-30 days)
  Self-reported depressive symptoms measured using the Beck Depression Inventory-II total score at pre and post-intervention. Potential range is 0-63, with higher scores represented worse functioning/outcomes.
Increase in mean levels of positive affect from baseline to study completion for individuals in the PT and PTPSS intervention groups | from baseline to study completion (approximately 21-30 days)
  Positive affect was self-reported using the Modified Differential Emotion Scale (MDES). Potential range is 0 to 40, with higher scores reflecting higher levels of assessed emotions.
Mean level Change in Savoring Beliefs from baseline to study completion for individuals in the PT and PTPSS intervention groups | from baseline to study completion (approximately 21-30 days)
  Savoring beliefs were self-reported using the Savoring Beliefs Inventory (SBI) total score and subscales. Potential range is 24 to 168, with higher scores reflecting better outcomes/higher savoring beliefs.
Mean level Increase in mindfulness from baseline to study completion for individuals in the PT and PTPSS intervention groups | from baseline to study completion (approximately 21-30 days)
  Self reported mindfulness on the Carolina Empirically-Derived Mindfulness Inventory. Total score and subscale scores. Potential range 32-160 with higher scores reflecting higher levels of mindfulness / better outcomes.
Mean level Increase in life satisfaction from baseline to study completion for individuals in the PT and PTPSS intervention groups | from baseline to study completion (approximately 21-30 days)
  Self-reported life satisfaction using the Brief Satisfaction with Life Scale. Potential range 5-35, with higher scores reflecting higher satisfaction with life / better outcome.
Mean level Increase in perceived social support for individuals in the PTPSS intervention group from baseline to study completion | from baseline to study completion (approximately 21-30 days)
  Self report using the Medical Outcomes Study (MOS) Social Support Survey. Range is 1 to 5. Mean score calculated, with higher levels indicating more social support / better outcome.

SECONDARY OUTCOMES:
Mean level Increase in self-esteem for individuals in the PT and PTPSS intervention groups from baseline to study completion | from baseline to study completion (approximately 21-30 days)
  self-reported self-esteem on the Rosenberg Self-Esteem Scale. Scores range from 0 to 30, with higher scores reflecting higher self-esteem / better outcomes
Mean level Increase in gratitude from baseline to study completion for individuals in the PT and PTPSS intervention groups | from baseline to study completion (approximately 21-30 days)
  Self-report of gratitude using the Gratitude Questionnaire (GQ-6). Scores range from 6 to 24, with higher scores reflecting higher levels of gratitude / better outcome.
mean level Decrease in physical health symptoms from baseline to study completion | from baseline to study completion (approximately 21-30 days)
  Self-reported response on the frequency of 9 physical health symptoms over the past month. Scores range from 7 to 63. Higher levels reflect more physical heath problems / worse outcome.
Mean level Improvement in sleep from baseline to study completion for individuals in the PT and PTPSS intervention groups | from baseline to study completion (approximately 21-30 days)
  self-report on sleep duration and quality using the Pittsburgh Sleep Quality Inventory. Scores range from 0 to 21 with higher scores reflecting worse quality sleep / worse outcome

OTHER OUTCOMES:
Mean Level Changes in cognitive style for individuals in the PT and PTPSS intervention groups | from baseline to study completion (approximately 21-30 days)
  Self report using the Cognitive Style Questionnaire (CSQ). Range of scores is 72 (most positive) to 360 (most negative), with higher scores reflecting a more negative cognitive style.
Changes in Attentional Bias for individuals in the PT and PTPSS intervention groups | from baseline to study completion (approximately 21-30 days)
  Attention bias is measured using a computerized dot probe task in which individuals view two emotion faces on a computer screen and then indicate using a key stroke where the cursor showed up after the emotion faces images were briefly displayed. A bias toward negative faces is determined when the amount of time it takes an individual to identify the cursor when it appears in place of the negative emotion face over collective trials is faster, on average over the course of the trials, than when the cursor replaces the happy emotion face.
Change in interpretation bias in individuals in the PT and PTPSS intervention groups | from baseline to study completion (approximately 21-30 days)
  Using the Ambiguous situation task, participants read short stories with unclear social situations, then rate multiple possible interpretations of the situation. The task measures interpretation bias by assessing whether an individual consistently chooses the more negative or positive interpretations across several scenarios.
Photograph content | Photos will be taken starting on Day 1 and uploaded each day over the course of the 21 day intervention
  Participants in the PT and PTPSS will upload photos for the research team. The photos will be judged by independent raters on aspecs such as subject matter, positive nature of the photos, and for other trends.

IPD SHARING:
Plan to Share IPD: No
When the participants were consented, they were not asked whether their data could be shared outside of the individuals on the research team. Given that they did not give their consent to have data shared outside the research team, we have chosen not to do so.

REFERENCES:
- [Background] McKee LG, Algoe SB, Faro AL, O'Leary JL, O'Neal CW. Picture This! Bringing joy into Focus and Developing Healthy Habits of Mind: Rationale, design, and implementation of a randomized control trial for young adults. Contemp Clin Trials Commun. 2019 Jun 29;15:100391. doi: 10.1016/j.conctc.2019.100391. eCollection 2019 Sep. PMID 31372571

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-12-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT07313696/Prot_SAP_ICF_000.pdf